CLINICAL TRIAL: NCT02996266
Title: Impact of Fever Prevention in Brain Injured Patients
Acronym: INTREPID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: C. R. Bard (Industry)
Collaborators: Yale University (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMD-1111
Record Dates: First submitted 2016-12-05; First posted 2016-12-19 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Fever; Ischemic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage
Keywords: Targeted Temperature Management
MeSH Terms: conditions — Fever; Ischemic Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage | interventions — Hypothermia, Induced; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fever Prevention (Experimental): Fever will be prevented using a surface targeted temperature management system
  Interventions: Device: Targeted Temperature Management
- Standard Care (Active Comparator): Standard care in which fever may spontaneously develop
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Targeted Temperature Management — Prophylactic normothermia
  Other Names: Arctic Sun 5000 Temperature Management System
  Arms: Fever Prevention
Other: Standard Care — No intervention to control temperature unless fever occurs
  Arms: Standard Care

SUMMARY:
This study will assess the impact of fever prevention on fever burden and short- and long-term neurologic outcomes in brain injured patients. Half of the subjects will undergo fever prevention using a targeted temperature management system and half of the subjects will be treated for fever should it develop.

DETAILED DESCRIPTION:
Multiple studies demonstrate that fever / elevated temperature is associated with poor outcomes in brain injured patients; however, there are no conclusive studies that demonstrate that fever prevention/controlled normothermia is associated with better outcomes. This study will be conducted to assess the impact of advanced temperature control to prevent fever in brain injured patients. The fever prevention group will use the Arctic Sun Temperature Management System and will be compared to standard care patients in whom fever may spontaneously develop. If fever develops in a patient in the standard care group, they will be treated with standard fever care measures according to a step-wise algorithm, consisting primarily of intermittent antipyretics (e.g., acetaminophen) and cooling blankets and, when necessary, advanced targeted temperature management devices.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted with a primary neurological diagnosis of ischemic stroke, intracerebral hemorrhage, or subarachnoid hemorrhage
2. Prior to onset of acute symptoms, was considered functionally independent (mRS 0-2)
3. Meets disease-specific criteria

Exclusion Criteria:

1. Fever (≥38°C) prior to study enrollment
2. Pre-existing neurological, psychiatric, or other condition that would confound neurological assessment or would make it difficult to accurately assess neurologic and/or functional outcome
3. Has a pre-morbid condition with poor likelihood of survival to 6 months
4. Has a pre-morbid mRS ≥3
5. Diagnosed with brain death
6. Is undergoing therapeutic hypothermia therapy
7. Has sustained neurological injury felt to be catastrophic with little chance of recovery
8. Has a skin condition in which the use of the ArcticGel Pads is contraindicated (i.e., skin that has signs of ulceration, burns, hives, or rash)
9. Has poor skin integrity or poor tissue perfusion
10. Participation in a concurrent investigational / interventional study (medical device or drug)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Greer, MD, MA, Principal Investigator — Boston University; Kevin N. Sheth, MD, Principal Investigator — Yale University
Locations (40):
- United States (28):
  - University of Southern California, Los Angeles, California
  - Stanford University Hospital, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Rush University, Chicago, Illinois
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - The University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York - Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Providence St Vincent Medical Center, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Erlanger Health System Baroness Hospital, Chattanooga, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Harborview Medical Center, Seattle, Washington
- Australia (2):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Technische Universitat Dresden, Dresden
  - Universitätsklinikum Jena, Jena
  - LMU München, Klinikum Großhadern, Munich
- South Korea (4):
  - Keimyung University Dongsan Hospital, Daegu
  - Asan Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greer DM, Helbok R, Badjatia N, Ko SB, Guanci MM, Sheth KN; INTREPID Study Group. Fever Prevention in Patients With Acute Vascular Brain Injury: The INTREPID Randomized Clinical Trial. JAMA. 2024 Nov 12;332(18):1525-1534. doi: 10.1001/jama.2024.14745. PMID 39320879
- [Derived] Greer DM, Ritter J, Helbok R, Badjatia N, Ko SB, Guanci M, Sheth KN. Impact of Fever Prevention in Brain-Injured Patients (INTREPID): Study Protocol for a Randomized Controlled Trial. Neurocrit Care. 2021 Oct;35(2):577-589. doi: 10.1007/s12028-021-01208-1. Epub 2021 Mar 24. PMID 33761119
- [Derived] Cronberg T, Greer DM, Lilja G, Moulaert V, Swindell P, Rossetti AO. Brain injury after cardiac arrest: from prognostication of comatose patients to rehabilitation. Lancet Neurol. 2020 Jul;19(7):611-622. doi: 10.1016/S1474-4422(20)30117-4. PMID 32562686

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects screen failed after signing consent (n=9):
  Disease-specific criteria (Not met) = 3 Fever at time of study = 1 Fever for more than one hour or one instance prior to study enrollment = 3 Fever at time of randomization = 1 Aneurysmal SAH confirmed within 24 hours of symptom onset = 1
Period: Overall Study
Arm/Group | Fever Prevention | Standard Care
Started | 339 | 338
Completed | 211 | 222
Not Completed | 128 | 116

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fever Prevention | Standard Care | Total
Number analyzed (Participants) | 339 | 338 | 677
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (13.22) | 60.4 (13.86) | 60.7 (13.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 168 | 345
  Male | 162 | 170 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 26 | 57
  Not Hispanic or Latino | 307 | 312 | 619
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 68 | 66 | 134
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 56 | 68 | 124
  White | 204 | 189 | 393
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 18 | 37
  South Korea | 55 | 57 | 112
  United States | 223 | 224 | 447
  Switzerland | 10 | 9 | 19
  Germany | 32 | 30 | 62
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Missing height and weight for 3 patients to calculate BMI.
  kg/m^2
    number analyzed (Participants) | 338 | 336 | 674
    (all) | 28.51 (6.829) | 28.60 (6.827) | 28.56 (6.823)
Clinical Diagnosis [Count of Participants; unit: Participants]
  Intracerebral Hemmorrhage (ICH) | 111 | 112 | 223
  Ischemic Stroke (IS) | 128 | 126 | 254
  Subarachnoid Hemorrhage (SAH) | 100 | 100 | 200
Baseline Severity [Count of Participants; unit: Participants] — Population: Missing severity for 1 patient
  Participants
    number analyzed (Participants) | 338 | 338 | 676
    High (NIHSS ≥17, ICH ≥3, or WFNS ≥IV) | 156 | 158 | 314
    Low (NIHSS <17, ICH ≤2, or WFNS ≤III) | 182 | 180 | 362

OUTCOME MEASURES:

1. Primary Outcome: Fever Burden
Description: Daily average fever burden (°C-hour)
Time Frame: Up to 14 days
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: °C-hour
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
°C-hour | 0.37 (0.961) | 0.73 (1.075)

2. Secondary Outcome: Primary Neurologic Outcome: Modified Rankin Scale Short-Term
Description: Modified Rankin Scale is a 6-category outcome measurement with 0 = no limitations, no symptoms and 6 = death.
Time Frame: 3-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mRS score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
mRS score | 3.7 (1.41) | 3.6 (1.43)

3. Secondary Outcome: Other Neurologic Outcomes: NIH Stroke Scale Short-Term
Description: NIH Stroke Scale is a systematic, quantitative assessment tool to measure stroke-related neurological deficit. Scores range from 0 to 42, with higher scores indicating worse outcome.
Time Frame: 3-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: NIHSS Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
NIHSS Score | 6.3 (6.30) | 6.7 (8.22)

4. Secondary Outcome: Other Neurologic Outcomes: Barthel Index Short-Term
Description: Barthel Index is an assessment of functional independence. Scores range from 0 to 100, with lower scores indicating worse outcome.
Time Frame: 3-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Barthel Index Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Barthel Index Score | 61.0 (36.35) | 59.6 (38.14)

5. Secondary Outcome: Other Neurologic Outcomes: Glasgow Outcome Scale Extended Short-Term
Description: Glasgow Outcome Scale assesses functional outcome after acute brain injury. Scores range from 1-8, with lower scores indicating worse outcome.
Time Frame: 3-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Glasgow Outcome Scale Extended Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Glasgow Outcome Scale Extended Score | 3.4 (1.98) | 3.6 (1.96)

6. Secondary Outcome: Other Neurologic Outcomes: Montreal Cognitive Assessment Short-Term
Description: Montreal Cognitive Assessment assesses for cognitive impairment. Scores range from 0-30, with lower scores indicating worse outcome.
Time Frame: 3-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: MOCA Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
MOCA Score | 17.6 (9.42) | 19.1 (9.62)

7. Secondary Outcome: Primary Neurologic Outcome: Modified Rankin Scale Mid-Term
Description: Modified Rankin Scale is a 6-category outcome measurement with 0 = no limitations, no symptoms and 6 = death.
Time Frame: 6-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mRS score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
mRS score | 3.5 (1.50) | 3.4 (1.60)

8. Secondary Outcome: Other Neurologic Outcomes: NIH Stroke Scale Mid-Term
Description: as for outcome 3
Time Frame: 6-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: NIHSS Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
NIHSS Score | 4.9 (5.05) | 5.6 (7.38)

9. Secondary Outcome: Other Neurologic Outcomes: Barthel Index Mid-Term
Description: as for outcome 4
Time Frame: 6-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Barthel Index Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Barthel Index Score | 65.4 (35.96) | 69.0 (35.26)

10. Secondary Outcome: Other Neurologic Outcomes: Glasgow Outcome Scale Extended Mid-Term
Description: as for outcome 5
Time Frame: 6-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Glasgow Outcome Scale Extended Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Glasgow Outcome Scale Extended Score | 3.6 (2.21) | 3.6 (2.22)

11. Secondary Outcome: Other Neurologic Outcomes: Montreal Cognitive Assessment Mid-Term
Description: as for outcome 6
Time Frame: 6-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: MOCA Score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
MOCA Score | 19.1 (8.93) | 20.0 (9.30)

12. Secondary Outcome: Primary Neurologic Outcome: Modified Rankin Scale Long-Term
Description: Modified Rankin Scale is a 6-category outcome measurement with 0 = no limitations, no symptoms and 6 = death.
Time Frame: 12-months post injury
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mRS score
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
mRS score | 3.5 (1.58) | 3.3 (1.64)

13. Secondary Outcome: Adverse Events
Description: An untoward medical occurrence, unintended disease or injury, or unanticipated complication
Time Frame: From date of randomization until hospital discharge, assessed up to 30 days
Population: As Treated
Measure: Number; unit: Adverse Events
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 331 | 336
Adverse Events
  Any Adverse Event during the Acute Phase | 933 | 764
  Any Adverse Event after the acute phase | 71 | 97
  Serious Adverse Event during the acute phase | 287 | 223
  Serious Adverse Event after the acute phase | 68 | 88

14. Secondary Outcome: Major Adverse Events
Description: MAEs defined as one of the following: pneumonia, sepsis, malignant cerebral edema, death
Time Frame: From date of randomization until end of study, assessed up to 12 months
Population: As Treated
Measure: Number; unit: Major Adverse Events
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 331 | 336
Major Adverse Events
  MAE through 3 months | 213 | 201
  MAE through 6 months | 228 | 227
  MAE through 12 months | 235 | 241

15. Secondary Outcome: Number of Participants With Infection
Description: Healthcare associated infection
Time Frame: From date of randomization until hospital discharge, assessed up to 30 days
Population: As Treated
Measure: Count of Participants; unit: Participants
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 331 | 336
Participants | 112 | 116

16. Secondary Outcome: Number of Subjects With Shivering
Description: Shivering greater than or equal to 1 on the Bedside Shivering Assessment Scale (BSAS). BSAS scores range from 0-3 with 0 indicating no shivering noted and 3 indicating severe shivering involving gross movements of the trunk and upper and lower extremities.
Time Frame: Up to 14 days
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Participants | 283 | 82

17. Other Pre Specified Outcome: Hospital Length of Stay
Description: Overall hospitalization duration
Time Frame: From date of randomization until hospital discharge, assessed up to 90 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Days | 25.3 (17.56) | 22.9 (16.04)

18. Other Pre Specified Outcome: ICU Length of Stay
Description: ICU Duration
Time Frame: From date of randomization until ICU discharge
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Hours | 335.096 (294.5559) | 312.949 (287.0900)

19. Other Pre Specified Outcome: Mortality
Description: Mortality
Time Frame: 7-day (or hospital discharge); 3-, 6-, and 12-months
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fever Prevention | Standard Care
Number analyzed (Participants) | 339 | 338
Participants | 75 | 77

ADVERSE EVENTS:
Time Frame: Data for all AEs was collected from randomization, up to 30 days. Data for Major Adverse Events was collected from randomization, up to 1 year.
Description: In this study, an MAE was defined as one of the following: Pneumonia, Sepsis, Malignant cerebral edema, or Death.
  All Adverse Events were analyzed using the As Treated (AT) population. This is the same as the Intent to Treat (ITT) population but based on the actual treatment received, not based on randomization, if there are patients who received the treatment other than that which they were randomized to.
Arm/Group | Fever Prevention | Standard Care
All-Cause Mortality (participants affected / at risk) | 75/339 | 77/338
Serious Adverse Events (participants affected / at risk) | 150/331 | 132/336
Other Adverse Events (participants affected / at risk) | 122/331 | 48/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fever Prevention (N=331) | Standard Care (N=336)
Brain Oedema (Nervous system disorders) | 27 | 29
Pneumonia (Infections and infestations) | 45 | 48
Urinary Tract Infection (Infections and infestations) | 31 | 1
Cerebral Vasoconstriction (Nervous system disorders) | 26 | 26
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 37 | 28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fever Prevention (N=331) | Standard Care (N=336)
Leukocytosis (Blood and lymphatic system disorders) | 18 | 7
Chills (General disorders) | 73 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 17 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT02996266/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT02996266/SAP_001.pdf